CLINICAL TRIAL: NCT06746051
Title: An Observational Study to Investigate Clinical Findings and Viral Load/Titer of Respiratory Syncytial Virus (RSV) Infection Over Time in Participants up to and Including 36 Months of Age
Brief Title: A Study to Investigate How Respiratory Syncytial Virus (RSV) Infection Develops and Changes Over Time in Pediatric Participants
Status: Completed | Type: Observational
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Other Study IDs: 2311T1492
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: RSV Infections
Keywords: Respiratory Syncytial Virus Infections; Lower Respiratory Tract Disease (LRTD)
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal swabs will be collected until the participant has no signs of RSV for 48 hours but not more than 10 days after RSV diagnosis via polymerase chain reaction (PCR).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Inpatients under 1 year of age: Participants <12 months of age who are PCR confirmed RSV positive and hospitalized for further evaluation of an acute respiratory tract illness will be actively enrolled with observational data collected for up to 21 days.
- Outpatients under 1 year of age: Participants <12 months of age who are PCR confirmed RSV positive and present in clinic for evaluation of an illness consistent with an acute respiratory tract infection will be actively enrolled with observational data collected for up to 21 days.
- Inpatients 1 to 3 years of age inclusive: Participants ≥ 12 months to ≤ 36 months of age who are PCR confirmed RSV positive and hospitalized for further evaluation of an acute respiratory tract illness will be actively enrolled with observational data collected for up to 21 days.
- Outpatients 1 to 3 years of age inclusive: Participants ≥ 12 months to ≤ 36 months of age who are PCR confirmed RSV positive and present in clinic for evaluation of an illness consistent with an acute respiratory tract infection will be actively enrolled with observational data collected for up to 21 days.

SUMMARY:
The primary purpose of this study is to observe how viral load and titer change over time in participants with RSV and how data from hospitalized participants compares with data from non-hospitalized participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant who is presenting within 5 days of onset of clinical signs at the time of informed consent.
* Participant is diagnosed with RSV within 5 days of sign onset.
* Participant's caregiver must be able to complete daily Observer Reported Outcomes (ObsROs) and collect nasal swabs

Key Exclusion Criteria:

* Participant is hospitalized for reasons other than RSV infection.
* Participant is considered by the PI to be immunocompromised, due to an underlying medical condition or medical therapy.
* Participant has or has had a confirmed respiratory infection with another clinically relevant viral/bacterial pathogen within 14 days of study enrollment.
* Participant underwent major surgery within 28 days prior to enrollment in the study or has planned major surgery within 15 days of expected study completion.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be enrolled at both inpatient and outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in RSV Viral Load Measurements | Day 1 to Day 21
  Viral load will be reported from results of quantitative reverse-transcription polymerase chain reaction (qRT-PCR).
Change From Baseline in RSV Viral Titer Measurements | Day 1 to Day 21
  Infectious viral titer will be reported from results of quantitative virus culture on adherent cells using a ViroSpot immunostaining readout.

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (2):
- United States (2):
  - SUNY Upstate Medical University, Syracuse, New York
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No